CLINICAL TRIAL: NCT04224584
Title: A Mechanism Based Proof of Concept Study of the Effects of Duloxetine in the Treatment of Patients With Osteoarthritic Knee Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kristian Kjær Petersen (Other)
Collaborators: CCBR, Aalborg (Unknown); Aalborg University Hospital (Other)
Responsible Party: Sponsor-Investigator, Kristian Kjær Petersen, Associate Professor, M.Sc., Ph.D., Aalborg University
Organization: Aalborg University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: DULKOA2019
Record Dates: First submitted 2020-01-06; First posted 2020-01-13 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duloxetine (Active Comparator): Duloxetine is a serotonin-norepinephrine reuptake inhibitor. Duloxetine will be administrated as follows: 20 mg/daily duloxetinefor 1 week, 40 mg/daily duloxetine for 1 week, 60 mg/daily duloxetine for 10 weeks, 40 mg/daily duloxetine for 1 week, 20 mg/daily duloxetine for 1 week.
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator): Placebo will be administrated for 14 weeks.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Duloxetine — Duloxetine will be administrated with a two weeks up titration followed by a 10 weeks full treatment (60 mg/daily) and finalized by a two weeks discontinuation.
  Arms: Duloxetine
Drug: Placebo oral tablet — Placebo will act as a control for duloxetine.
  Arms: Placebo

SUMMARY:
Background: Duloxetine provides an analgesic effect of patients with OA. The mode of action of duloxetine is partly believed to act through modulating the descending inhibitory pain pathways from the brainstem towards the spinal cord thereby dampening pain by gating the afferent pain signals from the periphery during their passage to the brain. This study aims to investigate if the analgesic effect of duloxetine is due to modulation of pain mechanisms.

Study Rationale: The present study will utilize a set of quantitative pain biomarkers developed to assess peripheral and central manifestations in OA and the influence of duloxetine on those manifestations.

Treatment: Patients will be randomized to one of two treatment sequences:

1. Sequence 1: 20 mg duloxetine QD for 1 week, 40 mg Duloxetine QD for 1 week, 60 mg duloxetine QD for 10 weeks, 40 mg duloxetine QD for 1 week, 20 mg duloxetine QD for 1 week, followed by 14 weeks of corresponding placebo
2. Sequence 2: 14 weeks of placebo followed by 20 mg Duloxetine QD for 1 week, 40 mg duloxetine QD for 1 week, 60 mg duloxetine QD for 10 weeks, 40 mg duloxetine QD for 1 week and 20 mg duloxetine QD for 1 week.

The two treatment periods of 14 weeks each are separated by a washout period of two weeks and include a two-week titration period.

Primary Objective: To assess the effect of 60 mg daily maintenance dose administration of Duloxetine for 10 weeks compared with placebo on pain mechanisms.

Sample Size Justification/Statistics: The sample size was calculated to 32 patients providing a power of 85% with a significant level of 0.05 to detect a group difference of 1 point in the change from baseline of the week 12 mean of 24-hour worst pain between duloxetine and placebo treatment.

Patient Selection: Up to 40 patients with osteoarthritic knee pain will be enrolled in this study in order to complete 32 patients.

Study sites:

Mech-Sense Aalborg University Hospital, DK-9000 Aalborg, Denmark Study Assessments: As the primary objective of this study is the assessment of which pain mechanisms are modulated by administration of the study drug, the primary endpoints will be Experimental Mechanism Based Pain Measures (EPMs) including 1) Pressure Pain Thresholds (PPTs), Temporal Summation, Conditioned Pain Modulation (CPM) and Offset Analgesia. In addition, efficacy will be evaluated using 1) pain severity (worst daily pain and night pain), 2) Pittsburgh Sleep Quality Index (PSQI), 3) Brief Pain Inventory (BPI), 4) Investigator and Patient Global Assessment of Changes (IGIC and PGAC), 5) Western Ontario and MacMaster (WOMAC) OA physical function, 6) PainDetect, and 7) Central Sensitization Index (CSI).

Safety: Discontinuation rates and Treatment Emergent Adverse Events (TEAEs). Key Inclusion/Exclusion Criteria: Males or females between 40 and 75 years of age, who are postmenopausal or using allowed contraception methods, and have a Body Mass Index (BMI) between 20-35 kg/m2 inclusive Patient with unilateral or bilateral OA of knee diagnosed according to the American College of Rheumatology (ACR) criteria based on clinical and radiographic evidence with pain severity equal to or higher than 5 on a Visual Analogue Scale (VAS) assessed as the worst pain within the last 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent and abide by the study restrictions.
2. Males and females between 40 and 75 years of age and body weight >40 kg and <150 kg with a body mass index (BMI) between 20-35 kg/m2 inclusive
3. Patients with osteoarthritic knee based on disease diagnostic criteria as presented in section; Inclusion Disease Criteria.
4. Self-reported pain intensities higher or equal to 5 cm on a 0-10 cm visual analog scale when asked to assess the worst pain within the last 24 hours
5. Have agreed to maintain the same activity level throughout the course of the study.
6. Knee pain for at least 14 days per month for the last three months before study entry.
7. Osteophytes (with radiographic evidence).
8. At least 1 of the following 3 conditions: Age >50, or morning stiffness <30 minutes, or crepitus.
9. Kellgren and Lawrence grade of I, II or III at the index knee. If the patient has had X-rays of the knee joints within the last year, which can confirm the diagnosis, they may be used. Otherwise, a new posterior-anterior view X-ray of both knees will be conducted by CCBR Aalborg.
10. Worst pain within the last 24-hour must be 5.0cm to 10.0cm (assessed on a 0-10 cm VAS scale anchored at 0cm: no pain and 10cm: worst pain imaginable) prior to enrolment.
11. Discontinued use of all analgesic medications (including over-the-counter [OTC] analgesics/ Non-Steroidal Anti-Inflammatory Drug (NSAID) at least three days prior to randomization (patients are allowed limited use of analgesic medications).

Exclusion Criteria:

1. Have a history of recurrent seizures other than febrile seizures.
2. Have a history of frequent and/or severe allergic reactions with multiple medications.
3. Patients with a current or recent history, as determined by the PI or his delegates, of severe, progressive, and/or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, psychiatric or cerebral disease which could interfere with the patient's participation in the study.
4. Moderate or great hepatic impairment. Retest of abnormal lab values is allowed once. If still abnormal, the patient will be excluded.
5. An alanine aminotransaminase (ALAT) higher than the Upper Limit of Normal (ULN) or explain by obesity
6. Have prior renal transplant, current renal dialysis or severe renal insufficiency (creatinine clearance of <30 mL/min), or serum creatinine laboratory value >1.5 times ULN, based on the reference ranges of the central laboratory.
7. Have uncontrolled hypertension (systolic blood pressure over 160 and diastolic blood pressure over 100)
8. Have active peptic ulcer, gastrointestinal (GI) bleeding or previous unexplained bleeding episodes
9. Have known inflammatory intestinal disease or gastrointestinal disease which might impact absorption
10. Patients with congestive heart failure (NYHA II-IV)
11. Bazett's corrected QT (QTcB) interval > 450 msec for men and > 470 msec for women
12. Patients with diabetes mellitus and documented atherosclerosis
13. Patients allergic to the active ingredient of duloxetine or one or more of the excipients
14. Pregnancy and breast feeding
15. Non-postmenopausal (defined as the absence of menstruation for at least 12 months and confirmed by assessing the follicle-stimulating hormone (FSH) level) and non-sterile females patients not using fertility control such as either birth control pills, hormonal or copper intrauterine device (IUD), vaginal ring, implant, transdermal release patch, or birth control depot injections
16. Patients with an active malignancy of any type or a history of malignancy within the last five years (except basal cell carcinoma of the skin that has been excised prior to study start)
17. Are taking any excluded medications (analgesic medications) that cannot be discontinued during the study period.
18. Patients in treatment with anticoagulants (with the exception of acetylsalicylic acid)
19. In treatment with a CYP1A2 inhibitors.
20. Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at Visit 1.
21. Have a history of substance abuse or dependence within the past year, excluding nicotine and caffeine
22. Patients at a high risk of infection (e.g. leg ulcers, indwelling urinary catheter and persistent or recurrent chest infections and patients who are permanently bed ridden or wheelchair bound)
23. Patients with a history of, or suspected, demyelinating disease of the central nervous system (e.g. multiple sclerosis or optic neuritis).
24. The investigator experiences that the volunteers do not fully understand the experimental pain procedures.
25. Investigator site personnel directly affiliated with this study and/or their immediate family. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
26. Patients on monoamine oxidase inhibitors (MAOIs), dopamine-antagonists, tricyclic antidepressants (TCAs), selective serotonin re-uptake inhibitors (SSRI)s or SNRIs, as well as use of the supplement St. John's Wort
27. Psychiatric diagnosis or symptoms (e.g. depression or anxiety) that in the opinion of the investigator could interfere with study procedures or participation evaluated using the Mini International Neuropsychiatric Interview (M.I.N.I.).
28. Has answered "yes" in the Columbia-Suicide Severity Rating Scale (C-SSRS) to suicidal ideation items 4 or 5, or any suicidal behaviour within six months before screening, at screening or at randomization visit, or has been hospitalized or treated for suicidal behaviour in the past five years before screening.
29. Patients are not allowed to donate blood or blood products during the study
30. Have secondary causes of arthritis of the knee including septic arthritis, inflammatory joint disease, articular fracture, major dysplasia or congenital abnormality, acromegaly, hemochromatosis, Wilson's disease, and primary osteochondromatosis.
31. Have had lower extremity surgery (including arthroscopy of the index knee) within 3 months prior to Visit 1 or have surgery planned of the index knee at any time.
32. Have had significant prior injury to the index knee within 12 months prior to Visit 1.
33. Use of lower extremity assistive devices other than a cane or knee brace (use of a 'shoe lift' is permitted). Are non-ambulatory or require the use of crutches or a walker. Use of a cane in the hand opposite the index knee is acceptable.
34. Has had a prior synovial fluid analysis showing a White Blood Cell (WBC) ≥2000mm3 that is indicative of a diagnosis other than OA at the index knee.
35. Have a confounding painful condition that may interfere with assessment of the index knee. (Knee pain should be the predominant pain. Mild OA of the hands is allowed, for instance).
36. Have any other musculoskeletal or arthritic condition that may affect the interpretation of the clinical efficacy and/or safety data or otherwise contraindicates participation in this clinical study (i.e., currently symptomatic fractures or any concurrent rheumatic diseases such as but not limited to fibromyalgia, rheumatoid arthritis, gout, pseudo-gout or Paget's disease and Reiter's syndrome are excluded).
37. Have used corticosteroids prior to baseline:

    1. Intra-articular injection of steroids to the index knee or into any other site than the index knee within the previous three months.
    2. Intra-muscular corticosteroid injections within the previous three months.
    3. Oral corticosteroids within the previous one month.
38. Have initiated or have changed to an established physiotherapy program within two weeks prior to Visit 2 or during the study period. An established physiotherapy program may be continued throughout the study period if unchanged in frequency and intensity.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold. | Difference between baseline (prior to treatment) compared with 10 weeks of 60 mg/daily duloxetine compared with placebo
  Assessment of pressure hyperalgesia. The Pressure Pain Threshold is assessed using a Somedic Handheld algometer (Somedic AB, Sösdala, Sweden). The Pressure Pain Threshold is assessed in kPa (kilo pascal).

CONTACTS AND LOCATIONS:
Locations (1):
- Mech-Sense, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ammitzboll N, Arendt-Nielsen L, Bertoli D, Brock C, Olesen AE, Kappel A, Drewes AM, Petersen KK. A mechanism-based proof of concept study on the effects of duloxetine in patients with painful knee osteoarthritis. Trials. 2021 Dec 27;22(1):958. doi: 10.1186/s13063-021-05941-y. PMID 34961547